CLINICAL TRIAL: NCT04779671
Title: Effects of the Fully Immersive Virtual Reality Cognitive Training Based on Leisure Activities for the Elderly With Mild Cognitive Impairment and Subjective Cognitive Decline.
Brief Title: Effects of the Fully Immersive VR Cognitive Training Based on Leisure Activities for the Elderly With MCI and SCD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202002283B0
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: MCI; SCD; Virtual Reality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental)
  Interventions: Behavioral: VR cognitive training
- control group (Active Comparator)
  Interventions: Behavioral: Traditional cognitive training

INTERVENTIONS:
Behavioral: VR cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  They will receive one immersive leisure-based VR cognitive training for 30 minutes. VR cognitive training receives four gardening activities.
  The cognitive elements including attention, working memory, processing speed, and executive function incorporated training.
  Arms: VR group
Behavioral: Traditional cognitive training — All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions.
  The control group is performing traditional cognitive training program.
  Arms: control group

SUMMARY:
Mild cognitive impairment (MCI) and subjective cognitive decline (SCD) are risk groups for dementia, and thus appropriate interventions are required. Cognitive training is a common intervention applied to the elderly with cognitive decline.

Cognitive training integrated into leisure activities can increase the training motivation of the elderly, while improving cognitive performance and daily functions. Virtual reality (VR) can simulate daily living situations, and it can be an effective intervention with cognitive training. Although a few studies have found immersive VR cognitive training can improve the cognitive function of the elderly with cognitive decline, these studies have shown inconsistent results. In addition, it is yet not clear the long-term effect of fully immersive VR cognitive training and its impact on daily function. Furthermore, for immersive VR cognitive training, there is still a lack of training programs that integrate into the context of leisure activities. This type of VR cognitive training could help the effectiveness of cognitive training to be transferred into daily functions.

DETAILED DESCRIPTION:
This study aims to (1) determine the feasibility and usability of immersive leisure-based VR cognitive training; (2) identify the intervention effects of immersive leisure-based VR cognitive training on cognitive function, daily function, and quality of life for elderly with MCI and SCD; (3) compare the intervention effects between elderly with MCI and SCD on outcome measures.

The investigators will recruit 30 elderly with MCI, 30 elderly with SCD, and 15 specialists for the feasibility and usability study. They will receive one immersive leisure-based VR cognitive training for 30 minutes. VR cognitive training receives four gardening activities. The cognitive elements including attention, working memory, processing speed, and executive function incorporated training. The investigators will use the Acceptance of the Virtual Reality (VR) Experience Questionnaire and System Usability Scales. For effectiveness study, the investigators will recruit 60 elderly with MCI and 70 elderly with SCD. Participants will be randomly assigned to VR group and control group. All participants will receive trainings for 60 minutes per day, two days per week for 16 sessions. The content of VR training is the same as before. The control group is performing traditional cognitive training program. The primary cognitive outcome measurements will include the Montreal Cognitive Assessment, Wechsler Memory Scale, Stroop test, and color trials test. Other outcomes will include measurements that evaluate the cognitive, daily functions, and quality of life of elderly with MCI and SCD. Participants will be assessed at baseline, after the intervention, and at 3-month follow-up. Repeated measures of analysis of variance (ANOVA) will be used to evaluate the changes in outcome measures at three different time points.

The investigators anticipate the VR training can facilitate cognitive function, daily function, and quality of life. The significance of this study is identifying the effect of immersive VR cognitive training based on leisure activities, and it is appropriate to provide this training for elderly with MCI and SCD. It could delay and prevent the progression to dementia and lead the field of technological assistance to new opportunities for training.

ELIGIBILITY:
MCI Inclusion Criteria:

* age range from 60 to 90 years
* self- or informant-reported memory or cognitive complaint.
* able to follow instruction
* MMSE score <26
* dose not have dementia.

SCD Inclusion Criteria:

* age range from 60 to 90 years;
* MMSE>=26;
* ECog-12 score >1;
* does not conform the standards of MCI and dementia .

Exclusion Criteria:

* dizziness or epilepsy history;
* neurological or other orthopedic diseases with neurological or other orthopedic diseases unstable physical condition of VR cognitive training;
* Recent psychiatric diagnosis, such as depression.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA) | baseline, posttest (around 12 weeks after baseline)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change scores of the Wechsler Memory Scale - Third Edition (WMS-III) | baseline, posttest (around 12 weeks after baseline)
  Several subtests of Wechsler Memory Scale - Third Edition (WMS-III) including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Stroop Color-Word Test | baseline, posttest (around 12 weeks after baseline)
  The Stroop Color-Word test assesses the abilities of selective attention, inhibition and executive function. The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. In both conditions, the number of colors correctly named within 45 seconds will be measured and the performance in the congruent condition will be compared with the incongruent condition.

SECONDARY OUTCOMES:
Change scores of the Wechsler Adult Intelligence Scale (WAIS) | baseline, posttest (around 12 weeks after baseline)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of the Everyday Cognition scales (ECog)-12 items | baseline, posttest (around 12 weeks after baseline)
  To detect cognitive and functional decline. The ECog shows promise as a useful tool for the measurement of general and domain-specific everyday functions in the elderly. There are six domains (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided Attention) in ECog. Lower scores represent a higher level of function in daily life.
Change scores of the Lawton Instrumental Activities of Daily Living Scale (IADL) | baseline, posttest (around 12 weeks after baseline)
  Assess activities of daily living. There are 8 domains of function measured with the Lawton IADL scale, including ability to use phone,shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications,and ability to handle finances. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent). For each category, circle the item description that most closely resembles the client's highest functional level (either 0 or 1).
Change scores of the WHOQOL-BREF Taiwan Version | baseline, posttest (around 12 weeks after baseline)
  Exploratory and confirmatory factor analyses revealed a four-factor (physical, psychological, social, and environmental) model. The internal consistency (Cronbach's α) coefficients ranged from 0.70 to 0.77 for the four domains. The test-retest reliability coefficients with intervals of 2 to 4 weeks ranged from 0.41 to 0.79 at item/facet level and 0.76 to 0.80 at domain level (all p < 0.01). Content validity coefficients were in the range of 0.53 to 0.78 for item-domain correlations and 0.51 to 0.64 for inter-domain correlations (all p < 0.01). The four domains of the brief form can explain 88% of the variance of the total QOL score and 60% of the variance of the Facet G score (measuring overall quality of life and general health).
Change scores of Geriatric Depression Scale (GDS) | baseline, posttest (around 12 weeks after baseline)
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.
Change scores of The Chinese Aging Well Profile (CAWP) | baseline, posttest (around 12 weeks after baseline)
  The 31-item Chinese Aging Well Profile comprised seven subscales-'physical', 'psychological', 'independence', 'learning & growth', 'material', 'environmental', and 'social' well-being.

CONTACTS AND LOCATIONS:
Overall Officials: I-Ching Chuan, Ph.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan